CLINICAL TRIAL: NCT05559424
Title: Head-to-head Comparison of Stent Geometry Obtained by Different Ballooning Techniques in Large Bifurcations Treated by Provisional Stenting
Brief Title: Comparison of Results Achieved by Different Ballooning Techniques in Bifurcation Stenting
Acronym: CRABBIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Burzotta, Principal investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 5053
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Heart Disease
Keywords: Provisional; OCT; kissing balloon; bifurcations
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Before enrollment start, the plausibility of the study hypothesis will be verified in an experimental pilot randomized investigation conducted n an ex-vivo beating heart animal model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POT/KISSING/POT (PKP) (Active Comparator): * SB rewiring is performed with the objective to cross "distal" stent struts (distal rewiring) through pullback technique.
  * KBI is performed using short non-compliant balloons (balloon of MV sized in a 1:1 ratio with distal MV reference diameter and SB balloon sized in a 1:1 ratio with SB reference diameter), with sequential followed by simultaneous inflation.
  * Final POT is performed at the same way as initial POT
  Interventions: Diagnostic Test: OCT
- POT/SIDE/POT (PSP) (Active Comparator): * SB rewiring is performed with the objective to cross "distal" stent struts (distal rewiring) through pullback technique.
  * SB dilatation is performed with a balloon sized 1:1 according to SB reference diameter.
  * Final POT is performed at the same way as initial POT.
  Interventions: Diagnostic Test: OCT

INTERVENTIONS:
Diagnostic Test: OCT — OCT will be used to assess results after intervention

SUMMARY:
Single-stent strategy with provisional approach represents the gold standard for percutaneous coronary intervention of bifurcation lesions, and, according to European Bifurcation Club, performing provisional approach presents two steps considered as mandatory: "crossover stenting" in main vessel (MV) and subsequent post-dilation or "POT" (proximal optimization technique). While consensus exists regarding these first two steps, the exact optimal following sequence in case of side branch (SB) jeopardize after main vessel stenting is still a matter of debate.

Actually, the two most used techniques in this setting are represented by the simultaneous inflation of two balloons located respectively in the MV and SB followed by a second POT (POT/kissing balloon/POT technique) and the isolated inflation of a balloon placed in the SB followed by a second POT (POT/SIDE/POT technique).

The objective of this study is to compare the configuration achieved with POT/KISS/POT (PKP) and POT/SIDE/POT (PSP), using the "cutting edge" high-resolution intracoronary imaging modality (Optical Coherence Tomography, OCT).

DETAILED DESCRIPTION:
A preclinical phase of the study (CRABBS-VHL) was performed in isolated porcine hearts comparing the two common side-branch (SB) optimization techniques after stent implantation in the main vessel (MV): proximal optimization technique (POT) + kissing balloon inflation + final POT (PKP arm) and POT + isolated balloon inflation + final POT (PSP arm).

A total of 30 PCIs were successfully performed. Baseline characteristics of treated bifurcations were similar between the two study arms. Minimum stent expansion at the distal main vessel (MV) segment was significantly lower with PSP as compared with PKP as assessed by both OCT and Micro-CT . Other significant findings included: higher stent eccentricity index at proximal MV with PSP, higher SB scaffolding length and lower malapposition (at bifurcation core and distal MV) with PKP.

These data need to be confirmed by further randomized studies in humans.

ELIGIBILITY:
Clinical inclusion criteria:

* Subject has coronary artery disease involving a bifurcation with evidence of myocardial ischemia, including patient with chronic coronary syndromes, unstable angina, or non-ST elevation-acute coronary syndromes (NSTE-ACS) hemodynamically stable.
* Subject is suitable to be treated by PCI according to operator's judgement or heart team decision.
* PCI planning includes provisional stenting and image guidance by OCT use.
* Patient is aged ≥ 18 years.
* Patient can provide written informed consent

Angiographic inclusion criteria:

- De novo coronary lesion involving the left main bifurcation, or a bifurcation lesion not located in the left main with large branches (distal MV reference diameter ≥ 3.5 mm and SB reference diameter ≥ 2.75 mm on visual estimation)

Clinical exclusion criteria:

* Acute coronary syndromes with ST-elevation (STE-ACS)
* Cardiogenic shock
* LVEF ≤ 30%
* Pregnancy
* Known severe thrombocytopaenia (platelet count < 50,000/mm3)
* eGFR ≤ 30 mL/min/m2 (Cockcroft-Gault)
* Contraindications to antiplatelet drugs/anticoagulant drugs
* Significant allergic reactions for contrast agent
* Women with pregnancy potential.

Angiographic exclusion criteria:

* Target chronic total occlusion
* Planned 2 stent-strategy
* Target bifurcation lesion has a previously implanted stent
* Target graft lesions
* Medina 0.0.1 target lesions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Stent expansion | Intra-procedural
  Minimum stent expansion

SECONDARY OUTCOMES:
Side branch ostial scaffolding length | Intra-procedural
  difference between maximal stent diameter at bifurcation core and distal reference diameter
Stent eccentricity index | Intra-procedural
  SEI = minimum stent diameter/maximum stent diameter
Stent complications | Intra-procedural
  Stent under-expansion
Additional treatment after OCT | Intra-procedural
  need of additional treatment after assessment of results by OCT
Stent malapposition | Intra-procedural
  Stent malapposition
Stent proximal edge dissection | Intra-procedural
  Stent proximal edge dissection
Tissue prolapse | Intra-procedural
  Tissue prolapse
Intracoronary thrombus | Intra-procedural
  Intracoronary thrombus
Side branch ostium dissection | Intra-procedural
  Side branch ostium dissection
Stent complicatons | Intra-procedural
  In-stent dissection

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Policlinico A. Gemelli. Università Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No